CLINICAL TRIAL: NCT07142213
Title: Effect and Mechanism of Combined Hepatectomy and Portal Vein Ligation Staged Hepatectomy (ALPPS) on Liver Regeneration in Patients With Hepatobiliary Malignancy
Brief Title: Effect and Mechanism of ALPPS Operation on Liver Regeneration
Status: Recruiting | Type: Observational
Sponsor: Haitao Zhao, MD (Other)
Responsible Party: Sponsor-Investigator, Haitao Zhao, MD, Deputy chief of liver surgery, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: K7100
Record Dates: First submitted 2025-01-13; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2024-12

CONDITIONS: Hepato Cellular Carcinoma (HCC); Hepatobiliary Cancers; Liver Cancer; Liver Regeneration
Keywords: liver regeneration; ALPPS; hepatectomy
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ALPPS group: Patietns who undergoing associating Liver Partition and Portal Vein Ligation for Staged Hepatectomy (ALPPS)
  Interventions: Procedure: ALPPS

INTERVENTIONS:
Procedure: ALPPS — In recent years, Associating Liver Partition and Portal Vein Ligation for Staged Hepatectomy (ALPPS) provides new hope for the solution of large/unresectable hepatobiliary malignancies. This technique promotes the rapid proliferation and regeneration of the remaining liver by separating the liver and ligation of the portal vein, so that the patients whose original liver function is not enough to tolerate large-scale liver resection can complete liver regeneration in a short time, so as to perform secondary resection. Compared with traditional two-stage hepatectomy, ALPPS significantly speeds up the rate of liver regeneration, shortens the waiting time for a second surgery, and provides a safer radical treatment for tumors in high-risk patients.

SUMMARY:
Hepatobiliary malignancies-principally hepatocellular carcinoma (HCC) and cholangiocarcinoma (CCA)-are highly aggressive and often diagnosed at advanced stages. Curative-intent liver resection remains the standard for resectable disease; however, postoperative outcomes depend on an adequate functional future liver remnant (FLR). Associating Liver Partition and Portal Vein Ligation for Staged Hepatectomy (ALPPS) induces rapid FLR hypertrophy and has expanded resection eligibility compared with conventional two-stage hepatectomy by shortening the interval to definitive resection.

Key uncertainties persist regarding the quality of ALPPS-induced regeneration and its relationship to long-term oncologic outcomes, including recurrence and metastasis. This observational study enrolls patients deemed suitable for ALPPS at Peking Union Medical College Hospital. Perioperative care follows institutional standards; no therapeutic procedures are altered for research purposes. The investigators will collect clinically available liver tissue and relevant medical data obtained during standard surgical care to characterize cellular and molecular programs of regeneration across the ALPPS stages.

High-throughput profiling-including single-cell and spatial transcriptomics-will be used to define cell-type composition, transcriptional states, and signaling pathways associated with regeneration. The primary objective is to describe cellular and gene-expression changes in regenerating liver induced by ALPPS. Secondary objectives include exploring associations between regenerative quality and short- and long-term clinical outcomes. Findings are expected to inform potential therapeutic targets and strategies to enhance safe regeneration and improve postoperative prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Patients aged 18 to 75 years
2. Diagnosis established: A diagnosis of hepatobiliary malignancy (including hepatocellular carcinoma and cholangiocarcinoma) was confirmed and evaluated as suitable for ALPPS surgery
3. Liver function status: preoperative Child-Pugh score A or B, MELD score ≤15, with sufficient liver function reserve for operation
4. Tumor characteristics: bilobal or complex tumors of the liver with large tumor areas requiring ALPPS to ensure adequate residual liver volume (FLR/TLV<30% or FLR/BW<0.5)
5. Preoperative assessment: Imaging showed that future liver residual (FLR) was insufficient to support standard hepatectomy, and liver volume must be increased by ALPPS
6. FLR enlargement: Postoperative assessment of FLR enlargement as expected (at least 30% enlargement or FLR/BW above 0.5) for a second procedure
7. No distant metastases: No unresectable extrahepatic metastases, except for resectable lung metastases

Exclusion Criteria:

1. Preoperative FLR insufficiency: Residual liver volume (FLR) did not increase sufficiently after the first step (<30% increase or FLR/BW <0.5) to be suitable for the second step
2. Extrahepatic metastasis: unresectable distant metastasis, such as extensive metastasis of bone, lung, etc
3. Severe liver disease: very poor liver function before surgery, Child-Pugh grade C or severe liver sclerosis during surgery (e.g. Metavir≥F3 or 30% or more hepatic steatosis)
4. Major comorbidities: Major illnesses such as severe cardiovascular disease, kidney failure, or respiratory failure that do not tolerate major surgery
5. Postoperative complications: Serious postoperative complications (such as liver failure, infection, etc.) after the first step are not suitable for the second step
6. Evaluation of adverse surgery: After the first procedure, FLR blood supply or function is abnormal, affecting liver regeneration
7. Pregnancy and lactation: pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with radiologically or pathologically confirmed hepatobiliary malignancies
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Residual liver volume | Time Frame: Day 7 (±2 days) and Day 14 (±2 days) after Stage-1 ALPPS; primary analysis uses the last assessment obtained prior to Stage-2 (up to Day 28).
  Residual liver volume of the future liver remnant (FLR) immediately before Stage-2 resection, quantified by contrast-enhanced CT-based 3D volumetry; reported in milliliters (mL) and as percent of standard liver volume (%SLV).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Please contact the research contact person and submit a reasonable research proposal at the time of application

REFERENCES:
- [Background] Wen Z, Jin Z, Xu B, Zhu H, Wang J, Chen W, Zhang J, Huang K, Lan Z, Meng B, Mao W, Zhu H, Zhang L, Lu T, Zeng J, Bao L, Lau WY, Guo Y. Hepatic artery restriction operation combined with ALPPS (HARO-ALPPS), a novel ALPPS procedure for the treatment of hepatocellular carcinoma with severe fibrosis: retrospective clinical cohort study. Int J Surg. 2024 Sep 1;110(9):5662-5671. doi: 10.1097/JS9.0000000000001679. PMID 38768472